CLINICAL TRIAL: NCT00571246
Title: The Use of Anticonvulsants for Treatment of Patients With Alcohol Dependence and Post Traumatic Stress Disorder
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 0705002634
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Alcohol Dependence; Post Traumatic Stress Disorder
Keywords: treatment; Lamotrigine; Topiramate; alcohol dependence; post traumatic stress disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Topiramate; Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Topiramate (Experimental): Participants will be randomized to topiramate (250mg)
  Interventions: Drug: Topiramate
- Lamotrigine (Experimental): Participants will be randomized to lamotrigine (250mg)
  Interventions: Drug: lamotrigine
- Placebo (Placebo Comparator): Participants will be randomized placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Topiramate — Participants are randomized to take Topiramate (250mg/day) 2 times a day
  Arms: Topiramate
Drug: lamotrigine — Participants are randomized to take Lamotrigine (250 mg/day) 2 times a day
  Arms: Lamotrigine
Other: Placebo — Participants are randomized to take placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy of topiramate (250mg) or lamotrigine (250mg) versus placebo in reducing alcohol consumption and decreasing symptoms of PTSD in patients with comorbid AD and PTSD.

DETAILED DESCRIPTION:
There is a high rate of comorbidity with alcohol dependence (AD) and post traumatic stress disorder (PTSD). The rates of PTSD among individuals with AD are at least twice as high as those in the general population. In addition, alcohol dependence is the most common comorbid condition in men with PTSD. Despite this, little is known about how to best treat individuals with comorbid AD and PTSD. The use of anticonvulsants represents a novel approach to treatment that may target symptoms of both AD and PTSD. Both Topiramate and Lamotrigine act on the GABAergic and glutamatergic systems. Topiramate has GABAergic effects by robustly increasing brain GABA, and antiglutamatergic effects by inhibiting glutamate function that might antagonize alcohol's rewarding effects in AD and could contribute to the regulating of reexperiencing and arousal symptoms in PTSD. Lamotrigine is a glutamate-inhibiting anticonvulsant that has shown efficacy in some dually diagnosed patients with alcohol dependence, and in patients with PTSD. Neither topiramate nor lamotrigine have been used to treat patients with comorbid PTSD and AD. Methods: Ninety men and women with a current diagnosis of AD and PTSD will be enrolled in a 16-week trial. They will be assigned, in a double-blind fashion, to either topiramate, lamotrigine or placebo. Significance: This project will be the first to compare anticonvulsants (topiramate and lamotrigine) to placebo as effective treatments for reducing alcohol consumption and PTSD symptoms in patients with AD and PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18-60 years old.
2. Current alcohol abuse or dependence
3. Current PTSD
4. Patients with current alcohol dependence, with at least one recent episode of heavy drinking (defined as 5 or more drinks per drinking episode) over the past 14 days, and during a consecutive 30-day period within the 90 days prior to baseline evaluation.
5. Individuals who are on a stable dose (no less than 2 weeks) of antidepressant medication.
6. Medically and neurologically healthy on the basis of history, physical examination, EKG, screening laboratories (CBC w/ differential, TSH, Free-T4, ASAT, ALAT, GGT, BUN, creatinine, calcium, phosphorous, magnesium, total protein, albumin, electrolytes, VDRL, urinalysis, beta-HCG)
7. For women, negative pregnancy test and use of acceptable method of contraception.

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Individuals with a current unstable medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology (LFT > 3 times normal, abnormal BUN and creatinine, and unmanaged hypertension with BP > 200/120) which in the opinion of the physician would preclude the patient from fully cooperating or be of potential harm during the course of the study (includes those with a history of glaucoma, prostatic hypertrophy, urethral obstruction, cerebral arteriosclerosis, pyloric stenosis).
3. Patients who meet current SCID criteria for a major Axis I diagnosis (Bipolar Disorders, Schizophrenia and Schizophrenia-type Disorders).
4. History of substance dependence (other than alcohol, tobacco or cannabis) by DSM-IV criteria in the last 90 days.
5. Individuals taking mood stabilizers and antipsychotic medications.
6. Individuals with a history of allergies to topiramate or lamotrigine.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
drinking - measured using the TLFB | 16 weeks
craving - measured using the OCDS | 16 weeks
PTSD symptoms - measured using the CAPS | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L Petrakis, MD, Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States